CLINICAL TRIAL: NCT02357108
Title: A Trial on Patient's Evaluation of a Physician Conveying Two Different Messages
Brief Title: Message: Study of Patients' Perception of Physician's Compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 2012-0113; NCI-2015-01419 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Cancer
Keywords: Supportive Care; treatment options; doctor's compassion
MeSH Terms: interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Video/Doctor Sequence 1 (Active Comparator): Participants watch two videos with varying video/doctor sequence and complete 3 surveys (one before the first video and one survey after each video)
  Interventions: Other: Video; Behavioral: Survey
- Group 2: Video/Doctor Sequence 2 (Active Comparator): Participants watch two videos with varying video/doctor sequence and complete 3 surveys (one before the first video and one survey after each video)
  Interventions: Other: Video; Behavioral: Survey
- Group 3: Video/Doctor Sequence 3 (Active Comparator): Participants watch two videos with varying video/doctor sequence and complete 3 surveys (one before the first video and one survey after each video)
  Interventions: Other: Video; Behavioral: Survey
- Group 4: Video/Doctor Sequence 4 (Active Comparator): Participants watch two videos with varying video/doctor sequence and complete 3 surveys (one before the first video and one survey after each video)
  Interventions: Other: Video; Behavioral: Survey

INTERVENTIONS:
Other: Video — Watch two short videos with a 4-minute interval between the two of them, estimate 8 minutes to watch both the videos.
Behavioral: Survey — One set of surveys before first video and one set after each video played, estimate total of 30 minutes for all surveys.
  Other Names: Survey Questionnaires; questionnaire

SUMMARY:
The goal of this study is to learn what types of conversations patients prefer to have with their doctor about treatment options and how patients view their doctor's compassion.

DETAILED DESCRIPTION:
If participant agree to take part in the study, basic information will be collected (such as date of birth, date of diagnosis, sex, and religion). Participant will also complete questionnaires about any symptoms they may be having, how hopeful they are, how they are accepting the disease, their trust in the medical profession, and how they like information to be delivered to them.

After completing the questionnaires, they will be randomly assigned (as the roll of dice) to one of 4 groups.

Regardless of which group they are in, they will watch 2 short videos that show actors portraying a doctor and patient having a conversation about treatment options in a clinical setting. Both videos will discuss the same material, but the order of the videos and the actors in the videos will be different for each group. Both videos are about 4 minutes long.

After watching each video, the participant will complete 3 questionnaires about the doctor in the video. It should take about 38 minutes to watch both videos and to complete all of the questionnaires.

After they have watched both videos, they will be asked to choose which doctor they preferred and to briefly explain the reasons why they chose that doctor.

Length of Study:

Participant will be off study after they have completed the last questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced cancer, defined as locally advanced, recurrent or metastatic disease
2. Patients treated as outpatients by the Supportive and Palliative Care team.
3. Age >/= 18 years-old
4. English speaking
5. Normal cognitive status as determined by the interviewer based on the ability to understand the nature of the study and consent process.

Exclusion Criteria:

1) Patients suffering from a severe psychiatric disorder or condition that would significantly interfere with study participation, as determined by the Principal Investigator or by the attending palliative care physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Participant's Rating of Physician's Compassion | Approximately 38 minutes for video viewing and surveys.
  Physician compassion tested using compassion data from the first video viewed by each patient as assessed by a Physician Compassion Assessment survey. Patient's rating of physician's compassion by using a 5-item tool consisting of five 0-10 numerical rating scales assessing five dimensions: warm-cold, pleasant-unpleasant, compassionate-distant, sensitive insensitive, caring-uncaring. The sum of the five scales will give a final score representing physician's compassion with a 0 to 50 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberson C. Tanco, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tanco K, Rhondali W, Perez-Cruz P, Tanzi S, Chisholm GB, Baile W, Frisbee-Hume S, Williams J, Masino C, Cantu H, Sisson A, Arthur J, Bruera E. Patient Perception of Physician Compassion After a More Optimistic vs a Less Optimistic Message: A Randomized Clinical Trial. JAMA Oncol. 2015 May;1(2):176-83. doi: 10.1001/jamaoncol.2014.297. PMID 26181019
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org